CLINICAL TRIAL: NCT01165151
Title: Improving Weight Loss Maintenance Through Alternatives Schedules of Treatment
Brief Title: Impact of Group Size in Weight Loss Interventions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK081607-01A1
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Weight Loss
Keywords: obesity; weight loss; group size
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Small group (Experimental): 10-member groups
  Interventions: Behavioral: behavioral weight loss program
- Large group (Active Comparator): 30-member groups
  Interventions: Behavioral: behavioral weight loss program

INTERVENTIONS:
Behavioral: behavioral weight loss program — weekly, group-based lifestyle weight loss program

SUMMARY:
The present study will assess whether the size of treatment groups (groups of 10 vs. 30 participants) affects short- and long-term weight loss. It is hypothesized that participants assigned to a small group will exhibit similar short-term and long-term weight losses (i.e., weight loss at months 6 and 12) as compared to those assigned to a large group.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 21 years-old)
* Health insurance coverage with Capital Health Plan (CHP)
* Body mass index BMI between 30-45 kg/m2

Exclusion Criteria:

* BMI is less than 30 kg/m2 or greater than 45 kg/m2
* Weight loss > 10 pounds in past 6 months
* Acute or chronic illnesses for which weight loss is contraindicated
* Unwilling or unable to give informed consent
* Unwilling to accept random assignment
* Unwilling or unable to travel to CHP clinic for assessments and groups
* Likely to relocate out of the area in the next 12 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
change in weight from baseline to month 12 | 12 months

SECONDARY OUTCOMES:
adherence to treatment protocol | 12 months
  number and proportion of treatment sessions attended

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States